CLINICAL TRIAL: NCT06158399
Title: A Single-arm Clinical Study of Azacitidine in Combination With R-CHOP (ARCHOP) for the Treatment of TP53-mutated Previously Untreated Diffuse Large B-cell Lymphoma
Brief Title: AZA Combined With RCHOP in P53-mutated DLBCL.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Collaborators: Jiangsu Provincial People's Hospital (Other); Sun Yat-sen University (Other); Chinese Academy of Medical Sciences (Other); Shanxi Province Cancer Hospital (Other)
Responsible Party: Principal Investigator, Bing, Xu, Principal Investigator, The First Affiliated Hospital of Xiamen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XMDYYYXYK-07
Record Dates: First submitted 2023-11-22; First posted 2023-12-06 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: DLBCL - Diffuse Large B Cell Lymphoma; TP53
MeSH Terms: conditions — Dendritic Cell Sarcoma, Interdigitating | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ARCHOP (Experimental): Azacitidine in combination with R-CHOP
  Interventions: Drug: Azacitidine in combination with R-CHOP

INTERVENTIONS:
Drug: Azacitidine in combination with R-CHOP — Specified dose on specified days:
  Azacitidine (A) 100mg subcutaneous d-1 to d-5 Rituximab (R) 375mg/m2 IV d0 Cyclophosphamide (C) 750mg/m2 IV d1 epirubicin (H) 75mg/m2 IV d1 or liposomal adriamycin (D) 25-30mg/m2 IV d1 Vincristine (O) 1.4mg/m2 (max 2mg) IV d1 Prednisone (P) 100mg orally d1-5

SUMMARY:
To evaluate the efficacy and adverse effects of Azacitidine in combination with R-CHOP (ARCHOP) for the treatment of TP53-mutated previously untreated Diffuse large B-cell lymphoma

DETAILED DESCRIPTION:
This is a Phase 2, open-label clinical trial study that aims to evaluate the efficacy (eg. Complete response, Overall Survival, Progression Free Survival) and adverse effects of Azacitidine in combination with R-CHOP (ARCHOP) for the treatment of TP53-mutated previously untreated Diffuse large B-cell lymphoma

ELIGIBILITY:
Inclusion Criteria:

(1)18-70 years old; 2) New-onset TP53 mutant DLBCL; 3) ECOG 0-2; 4) LVEF >45%; 5) HBV-positive serology (occult carriers: anti-HBeAg +, HbsAg-, anti-HBsAg +/-) only if HBV-DNA test is negative before enrollment; (6) Liver function: serum bilirubin ≤ 2.0 × ULN, serum ALT and AST ≤ 2.5 × ULN. Renal function: serum Cr ≤ 2.0 × ULN; (unless due to lymphoma); 7) Life expectancy ≥ 6 months; 8) Informed consent.

Exclusion Criteria:

1. Primary and secondary central DLBCL;
2. HIV-positive patients and or HCV active infection; (3) Clinically significant secondary cardiovascular disease;

4) Combined hypoxemia severe chronic obstructive pulmonary disease; 5) Active bacterial, fungal, and, or viral infections not controlled by systemic therapy; 6) Apart from cured basal cell carcinoma of the skin or cervical cancer in situ or early prostate cancer not requiring systemic therapy or early breast cancer requiring only surgery alone. Within the last 3 years or concurrently with other malignant tumors; 7) Known hypersensitivity or allergic reaction to antibodies or proteins of the murine family

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2023-11-22 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Complete remission rate (CR) | Up to 36 months
  CR is evaluated according to the Lugano criteria for lymphoma response.

SECONDARY OUTCOMES:
Partial remission rate (PR) | Up to 36 months
  PR is evaluated according to the Lugano criteria for lymphoma response.
Overall response rate (ORR) | Up to 36 months
  Percentage of participants with best overall response of partial response (PR) and complete response (CR), using the Lugano criteria.
Progression Free Survival (PFS) | Up to 36 months
  The Kaplan-Meier method will be used to estimate the rate of PFS. PFS was defined as the time from the date of treatment initiation until the date of the first documented day of disease progression or relapse, using 2014 Lugano criteria, or death from any cause, whichever occurred first.

CONTACTS AND LOCATIONS:
Overall Officials: Bing Xu, Principal Investigator — The First Aiffiliated hosptical of xiamen University
Locations (1):
- Bing Xu, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No